CLINICAL TRIAL: NCT05482880
Title: Decisional Conflicts, Health-related Quality of Life and Satisfaction With Care in High-risk Cutaneous Squamous Cell Carcinoma in the Head-neck Region: Validated Questionnaires
Brief Title: Decisional Conflicts, Health-related QoL and Satisfaction With Care in High-risk cSCC in the Head-neck Region
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2018-2918-A-2
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Cutaneous Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinomas; Squamous Cell Carcinoma of Head and Neck; Squamous Cell Carcinoma of the Skin; Squamous Cell Carcinoma of the Head and Neck; Skin Cancer; High-Risk Cancer; Quality of Life; Satisfaction, Patient
Keywords: High-risk cutaneous squamous cell carcinoma; Health-related quality of life; Decisional conflicts; Satisfaction with care; Head-neck region; Multidisciplinary care
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Skin Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- head-neck cutaneous Squamous cell carcinomas: Patients with high risk cutaneous squamous cell carcinoma of the head-neck area receiving regular, multidisciplinary care.
  Interventions: Other: Regular care with additionally administration of questionnaires

INTERVENTIONS:
Other: Regular care with additionally administration of questionnaires — Patients receiving regular care. In addition, validated questionnaires are administered at two measurement points:
  1. after the multidisciplinary consultation, a baseline questionnaire*, the decision conflict scale and the EQ-5D-5L questionnaire are administered by phone.
  2. 1 month after completion of the treatment program (care pathway) the EQ-5D-5L, the BaSQoL and the EORTC IN-PATSAT32 questionnaires will be administered by phone.
  Completing the questionnaires takes about 30 minutes each time.
  *Baseline questionnaire: gender, age, marital status, education level, World Health Organization (WHO) performance status, presence of informal care, stage and treatment of cSCC, history of skin cancer, presence of current other skin cancer, and average travel time to hospital.

SUMMARY:
Patient reported outcomes in patients with high-risk cutaneous squamous cell carcinoma in the head-neck region are an important part of the complex care for these patients. Health-related quality of life, decision conflicts in the choice of treatment and satisfaction with care have not yet been sufficiently studied in this patient group.

DETAILED DESCRIPTION:
Cutaneous squamous cell carcinoma (cSCC) is the second most common form of skin cancer worldwide after basal cell carcinoma. It involves approximately 20% of all cutaneous malignancies and its incidence is still increasing. In 2020, nearly 15,000 cSCCs were reported in the Netherlands, of which approximately 50% concerned patients aged 75 years or older. UV radiation is the main risk factor for development of a cSCC, therefore the majority of cSCCs are localized to the sun-exposed skin in the head-neck region. cSCCs have a metastatic rate of 2.6-5% and recurrence rate of 1.9-3.7%, with rates increasing in high-risk cSCCs. The increasing incidence, advanced age, the (often) high-risk localization in the head-neck area (given functional and cosmetic importance) and the possible high risk of metastasis result in complex care, especially in stage T2 to T4 cSCCs, also known as high-risk cSCCs.

Patient-reported outcomes and health related quality of life (HRQoL) are important outcomes in the care for high-risk cSCCs in the head-neck region (HNcSCCs). Previous research is limited regarding the impact of cSCCs on QoL in patients with high-risk HNcSCCs , as is research on decision conflicts in the choice of treatment. The PROFILES registry (Arts, 2019) investigated QoL and satisfaction with care in 215 patients with keratinocyte carcinomas in the head-neck region. However, the majority of the patients had basal cell carcinoma (81%); only 23 patients had cSCC. Besides, no distinction was made in high or low risk cSCC. Finally, quality of life and patient satisfaction questionnaires were not administered until at least one year after diagnosis.

Other studies of QoL in cSCC patients do not distinguish stage and/or location of the tumor, involve small study populations, or only use oncological questionnaires rather than disease-specific questionnaires.

In conclusion, there is little scientific research on health related quality of life, decision conflicts in the choice of treatment and satisfaction with care in specific patients with high-risk HNcSCCs.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with a cutaneous squamous cell carcinoma located in the head-neck area (including patients with metastatic or recurrence disease)
* requiring a multidisciplinary approach
* assessed at the department of dermatology of Maastricht UMC+ or Radboud UMC OR discussed in the multidisciplinary consultation in Maastricht UMC+ or Radboud UMC
* and for which treatment of the tumor (primary tumor or metastatic/recurrence) takes places in the Maastricht UMC+ of Radboud UMC
* willing to participate voluntarily in the study

Exclusion Criteria:

* patients younger than 18 years
* patients with inadequate understanding of the Dutch language
* patients with cognitive impairment or otherwise unable to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected by the treating physicians from multidisciplinary consultation in the secondary/tertiary centers Maastricht UMC+ and Radboud UMC.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | At the start (before treatment) of the care pathway.
  Decisional conflicts expressed as mean total and domain scores on the Decisional Conflict Scale (DCS) questionnaire.
  The DCS questionnaire consist of 16 items related to decision conflicts. Items are given a score value of 0 (strongly agree), 1 (agree), 2 (neither agree or disagree), 3 (disagree) and 4 (strongly disagree). The total score can be calculated by summarize all scores, dividing by 16 and then multiplying by 25. The total score ranges from 0 to 100. A higher score correlates with a higher decisional conflict.
  The 5 domain subscores are: uncertainty (3 items), informed (3 items), values clarity (3 items), support (3 items) and effective decision (4 items). The subscores can be calculated by summarize the (3 or 4) items, dividing by the number of items (3 or 4) and then multiplying by 25. The subscores range from 0 to 100 where a higher score correlates with a higher decisional conflict.
Health-related quality of life | At the start (before treatment) of the care pathway.
  Health-related quality of life (HRQoL) expressed as mean total/domain scores on the EuroQol five-dimensional (5D) five-level (5L) (EQ-5D-5L) questionnaire.
  The EQ-5D-5L consist of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 response levels (no, slight, moderate, severe or extreme problems) resp. coded from 1 to 5. The EuroQol-visual analogue scale records the overall health on a vertical visual analogue scale (0 to 100). Example: a response of 77 is coded 77. A higher score indicates a better health status).
Health-related quality of life | At 1 month after completion of the care pathway.
  Health-related quality of life (HRQoL) expressed as mean total/domain scores on the EuroQol five-dimensional (5D) five-level (5L) (EQ-5D-5L) questionnaire.
  The EQ-5D-5L consist of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 response levels (no, slight, moderate, severe or extreme problems) resp. coded from 1 to 5. The EuroQol-visual analogue scale records the overall health on a vertical visual analogue scale (0 to 100). Example: a response of 77 is coded 77. A higher score indicates a better health status).
Health-related quality of life | At 1 month after completion of the care pathway.
  HRQoL expressed as mean total/domain scores on the Basal and Squamous Cell Carcinoma QoL (BaSQoL) questionnaire.
  The BaSQoL consist of 5 scales: behaviour, diagnosis/treatment, worries, appearance and other people. Items are scored: 0 (not at all), 1 (a little), 2 (quite a bit), 3 (very much). An average score per scale will be calculated (the sum of all scores within one scale, divided by the number of items) resulting in a scale score of 0 to 3. A higher score indicates a higher influence of skin cancer on daily life.
Satisfaction with care | Once during the care pathway: 1 month after completion of the care pathway.
  Satisfaction with care expressed as mean total and domain scores on the EORTC IN-PATSAT32 (patient satisfaction) questionnaire.
  The EORTC IN-PATSAT32 is composed of 11 multi-item scales (including doctors' and nurses' interpersonal skills, technical skills, information provision and availability, and other hospital personnel kindness/helpfulness and information giving, waiting time and access) and 3 single item scales (including exchange of information, comfort/cleanliness and general satisfaction). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a high level of satisfaction with care.

SECONDARY OUTCOMES:
Difference in decisional conflict outcomes between centers | At the start (before treatment) of the care pathway.
  Differences in decisional conflict outcome measures (primary outcome 1) between Maastricht University Medical Center+ and Radboud University Medical Center, expressed as mean total/domain scores on the Decisional Conflict Scale (DCS) questionnaire.
  The DCS questionnaire consist of 16 items related to decision conflicts. Items are given a score value of 0 (strongly agree), 1 (agree), 2 (neither agree or disagree), 3 (disagree) and 4 (strongly disagree). The total score can be calculated by summarize all scores, dividing by 16 and multiplying by 25 (total score range 0-100). A higher score correlates with a higher decisional conflict. The subscores are: uncertainty (3 items), informed (3 items), values clarity (3 items), support (3 items) and effective decision (4 items). The subscores can be calculated by summarize the items, dividing by the number of items and multiplying by 25. The subscores range from 0-100; a higher score correlates with a higher decisional conflict.
Difference in health-related quality of life outcomes between centers | At the start (before treatment) of the care pathway.
  Differences in health-related quality of life outcome measures (primary outcome 2) between Maastricht University Medical Center+ and Radboud University Medical Center. Health-related quality of life (HRQoL) expressed as mean total/domain scores on the EuroQol five-dimensional (5D) five-level (5L) (EQ-5D-5L) questionnaire.
  The EQ-5D-5L consist of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 response levels (no, slight, moderate, severe or extreme problems) resp. coded from 1 to 5. The EuroQol-visual analogue scale records the overall health on a vertical visual analogue scale (0 to 100). Example: a response of 77 is coded 77. A higher score indicates a better health status).
Difference in health-related quality of life outcomes between centers | At 1 month after completion of the care pathway.
  Differences in health-related quality of life outcome measures (primary outcome 3) between Maastricht University Medical Center+ and Radboud University Medical Center. Health-related quality of life (HRQoL) expressed as mean total/domain scores on the EuroQol five-dimensional (5D) five-level (5L) (EQ-5D-5L) questionnaire.
  The EQ-5D-5L consist of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 response levels (no, slight, moderate, severe or extreme problems) resp. coded from 1 to 5. The EuroQol-visual analogue scale records the overall health on a vertical visual analogue scale (0 to 100). Example: a response of 77 is coded 77. A higher score indicates a better health status).
Difference in health-related quality of life outcomes between centers | At 1 month after completion of the care pathway.
  Differences in health-related quality of life outcome measures (primary outcome 4) between Maastricht University Medical Center+ and Radboud University Medical Center. HRQoL expressed as mean total/domain scores on the Basal and Squamous Cell Carcinoma QoL (BaSQoL) questionnaire.
  The BaSQoL consist of 5 scales: behaviour, diagnosis/treatment, worries, appearance and other people. Items are scored: 0 (not at all), 1 (a little), 2 (quite a bit), 3 (very much). An average score per scale will be calculated (the sum of all scores within one scale, divided by the number of items) resulting in a scale score of 0 to 3. A higher score indicates a higher influence of skin cancer on daily life.
Difference in satisfaction with care outcomes between centers | At 1 month after completion of the care pathway.
  Differences in satisfaction with care outcome measures (primary outcome 5) between Maastricht University Medical Center+ and Radboud University Medical Center. Satisfaction with care expressed as mean total and domain scores on the EORTC IN-PATSAT32 (patient satisfaction) questionnaire.
  The EORTC IN-PATSAT32 is composed of 11 multi-item scales (including doctors' and nurses' interpersonal skills, technical skills, information provision and availability, and other hospital personnel kindness/helpfulness and information giving, waiting time and access) and 3 single item scales (including exchange of information, comfort/cleanliness and general satisfaction). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a high level of satisfaction with care.
Change from baseline health-related quality of life after treatment | Twice during the care pathway: at the start (before treatment) and 1 month after completion of the care pathway.
  The difference in HRQoL before and after treatment, expressed by mean total and domain scores on the EQ-5D-5L questionnaire.
  The EQ-5D-5L consist of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 response levels (no, slight, moderate, severe or extreme problems) resp. coded from 1 to 5. The EuroQol-visual analogue scale records the overall health on a vertical visual analogue scale (0 to 100). Example: a response of 77 is coded 77. A higher score indicates a better health status).

CONTACTS AND LOCATIONS:
Overall Officials: K Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud UMC, Nijmegen, Gelderland
  - Maastricht University Medical Center +, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stratigos AJ, Garbe C, Dessinioti C, Lebbe C, Bataille V, Bastholt L, Dreno B, Fargnoli MC, Forsea AM, Frenard C, Harwood CAlpha, Hauschild A, Hoeller C, Kandolf-Sekulovic L, Kaufmann R, Kelleners-Smeets NW, Malvehy J, Del Marmol V, Middleton MR, Moreno-Ramirez D, Pellecani G, Peris K, Saiag P, van den Beuken-van Everdingen MHJ, Vieira R, Zalaudek I, Eggermont AMM, Grob JJ; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO) and the European Organization for Research and Treatment of Cancer (EORTC). European interdisciplinary guideline on invasive squamous cell carcinoma of the skin: Part 1. epidemiology, diagnostics and prevention. Eur J Cancer. 2020 Mar;128:60-82. doi: 10.1016/j.ejca.2020.01.007. Epub 2020 Feb 26. PMID 32113941
- [Background] Stratigos AJ, Garbe C, Dessinioti C, Lebbe C, Bataille V, Bastholt L, Dreno B, Concetta Fargnoli M, Forsea AM, Frenard C, Harwood CA, Hauschild A, Hoeller C, Kandolf-Sekulovic L, Kaufmann R, Kelleners-Smeets NWJ, Malvehy J, Del Marmol V, Middleton MR, Moreno-Ramirez D, Pellecani G, Peris K, Saiag P, van den Beuken-van Everdingen MHJ, Vieira R, Zalaudek I, Eggermont AMM, Grob JJ; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO) and the European Organization for Research and Treatment of Cancer (EORTC). European interdisciplinary guideline on invasive squamous cell carcinoma of the skin: Part 2. Treatment. Eur J Cancer. 2020 Mar;128:83-102. doi: 10.1016/j.ejca.2020.01.008. Epub 2020 Feb 26. PMID 32113942
- [Background] Kallini JR, Hamed N, Khachemoune A. Squamous cell carcinoma of the skin: epidemiology, classification, management, and novel trends. Int J Dermatol. 2015 Feb;54(2):130-40. doi: 10.1111/ijd.12553. Epub 2014 Nov 27. PMID 25428226
- [Background] Que SKT, Zwald FO, Schmults CD. Cutaneous squamous cell carcinoma: Incidence, risk factors, diagnosis, and staging. J Am Acad Dermatol. 2018 Feb;78(2):237-247. doi: 10.1016/j.jaad.2017.08.059. PMID 29332704
- [Background] Mourouzis C, Boynton A, Grant J, Umar T, Wilson A, Macpheson D, Pratt C. Cutaneous head and neck SCCs and risk of nodal metastasis - UK experience. J Craniomaxillofac Surg. 2009 Dec;37(8):443-7. doi: 10.1016/j.jcms.2009.07.007. Epub 2009 Aug 27. PMID 19713116
- [Background] Brantsch KD, Meisner C, Schonfisch B, Trilling B, Wehner-Caroli J, Rocken M, Breuninger H. Analysis of risk factors determining prognosis of cutaneous squamous-cell carcinoma: a prospective study. Lancet Oncol. 2008 Aug;9(8):713-20. doi: 10.1016/S1470-2045(08)70178-5. Epub 2008 Jul 9. PMID 18617440
- [Background] Brougham ND, Dennett ER, Cameron R, Tan ST. The incidence of metastasis from cutaneous squamous cell carcinoma and the impact of its risk factors. J Surg Oncol. 2012 Dec;106(7):811-5. doi: 10.1002/jso.23155. Epub 2012 May 16. PMID 22592943
- [Background] Schmults CD, Karia PS, Carter JB, Han J, Qureshi AA. Factors predictive of recurrence and death from cutaneous squamous cell carcinoma: a 10-year, single-institution cohort study. JAMA Dermatol. 2013 May;149(5):541-7. doi: 10.1001/jamadermatol.2013.2139. PMID 23677079
- [Background] van Egmond S, Wakkee M, Droger M, Bastiaens MT, van Rengen A, de Roos KP, Nijsten T, Lugtenberg M. Needs and preferences of patients regarding basal cell carcinoma and cutaneous squamous cell carcinoma care: a qualitative focus group study. Br J Dermatol. 2019 Jan;180(1):122-129. doi: 10.1111/bjd.16900. Epub 2018 Sep 23. PMID 29927480
- [Background] Arts LPJ, Waalboer-Spuij R, de Roos KP, Thissen MRTM, Scheijmans LJ, Aarts MJ, Oerlemans S, Lybeert MLM, Louwman MWJ. Health-Related Quality of Life, Satisfaction with Care, and Cosmetic Results in Relation to Treatment among Patients with Keratinocyte Cancer in the Head and Neck Area: Results from the PROFILES Registry. Dermatology. 2020;236(2):133-142. doi: 10.1159/000502033. Epub 2019 Aug 21. PMID 31434078
- [Background] Chren MM, Sahay AP, Bertenthal DS, Sen S, Landefeld CS. Quality-of-life outcomes of treatments for cutaneous basal cell carcinoma and squamous cell carcinoma. J Invest Dermatol. 2007 Jun;127(6):1351-7. doi: 10.1038/sj.jid.5700740. Epub 2007 Feb 15. PMID 17301830
- [Background] Wang AY, Palme CE, Wang JT, Morgan GJ, Gebski V, Gilchrist J, Veness MJ. Quality of life assessment in patients treated for metastatic cutaneous squamous cell carcinoma of the head and neck. J Laryngol Otol. 2013 Jul;127 Suppl 2:S39-47. doi: 10.1017/S0022215113000303. Epub 2013 Mar 5. PMID 23458083
- [Background] Abedini R, Nasimi M, Noormohammad Pour P, Moghtadaie A, Tohidinik HR. Quality of Life in Patients with Non-melanoma Skin Cancer: Implications for Healthcare Education Services and Supports. J Cancer Educ. 2019 Aug;34(4):755-759. doi: 10.1007/s13187-018-1368-y. PMID 29705894